CLINICAL TRIAL: NCT06641245
Title: PREconception Folic Acid Clinical Efficacy (PREFACE) Trial
Acronym: PREFACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Crystal Karakochuk, Associate Professor, Human Nutrition, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H24-01716; UBC CREB H24-01716 (Other: The University of British Columbia (UBC) Clinical Research Ethics Board (CREB))
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Folate; Folate Bioavailability; Clinical Trials; Pregnancy
Keywords: Folic acid; Folate; Methylfolate; 5-MTHF; RBC Folate; Placental Growth Factor
MeSH Terms: interventions — Folic Acid; 5-methyltetrahydrofolate

STUDY DESIGN:
Intervention Model Description: A double-blind randomized non-inferiority trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5MTHF (Experimental): 5MTHF
  Interventions: Dietary Supplement: 5-MTHF (5-methyltetrahydrofolate)
- Synthetic folic acid (Active Comparator): Folic acid
  Interventions: Dietary Supplement: Folic Acid

INTERVENTIONS:
Dietary Supplement: Folic Acid — folic acid (0.6 mg)
  Arms: Synthetic folic acid
Dietary Supplement: 5-MTHF (5-methyltetrahydrofolate) — 0.625 mg/d (6S)-5-MTHF
  Arms: 5MTHF

SUMMARY:
A study to help understand what forms of folic acid are most effective to increase folate status during pregnancy for the best protection against neural tube defects

DETAILED DESCRIPTION:
A multisite randomized controlled trial to determine whether supplementation with (6S)-5-methyltetrahydrofolic acid (5-MTHF) is at least as effective as synthetic folic acid in increasing maternal folate status for protection against neural tube defects (NTDs).

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant females who are:
* Currently trying to become pregnant;
* Aged 19-42 years;
* Low risk for an NTD-affected pregnancy

Exclusion Criteria:

* Trying to conceive for ≥6 months (as ~90% of pregnancies occur after 6 months of trying);
* Diagnosed ovulatory disorders (polycystic ovary syndrome, endometriosis, or menstrual irregularity);
* More than 2 miscarriages in the past year;
* Undergoing fertility assistance (including current IVF or intrauterine insemination);
* Pre-existing medical condition known to impact maternal folate status (malabsorptive and inflammatory bowel diseases, active celiac disease, gastric bypass surgery, type 1 or 2 diabetes mellitus);
* Lifestyle factors known to impact maternal folate status (current smoking, >6 alcoholic drinks per week, recreational drug use);
* On the female or male side of those trying to conceive: personal NTD history, previous NTD-affected pregnancy, or personal or family history of other folate sensitive congenital anomalies;
* Use of folate-inhibiting medications (Chloramphenicol, Methotrexate, Metformin, Sulfasalazine, Phenobarbital, Phenytoin, Primidone, Triamterene, Barbiturates).

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 272 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
RBC folate | At 6 (± 2) wks gestation (approximate time of neural tube closure)
  •Maternal RBC folate concentrations (nmol/L)

SECONDARY OUTCOMES:
Maternal plasma placental growth factor (pg/mL) | At 18 (± 1) and 30 (± 1) wks gestation
  A novel biomarker with increasing use in clinical practice due to a discriminatory capacity for fetal growth restriction vs a small, but healthy fetus

OTHER OUTCOMES:
Human milk total folate concentrations | At 4 weeks postpartum
  Unmetabolized folic acid, reduced folate forms (nmol/L), and folate binding protein

CONTACTS AND LOCATIONS:
Overall Officials: Crystal D Karakochuk, PhD, Principal Investigator — The University of British Columbia; Kelsey M Cochrane, PhD, Principal Investigator — University of Saskatchewan

IPD SHARING:
Plan to Share IPD: No